# Title: Calcium Channel Blockade in Primary Aldosteronism Detailed Protocol

# NCT04179019

**Date of IRB Approval & Document Version: 1/9/2020** 

# I. BACKGROUND AND SIGNIFICANCE

Primary aldosteronism is the most common cause of secondary hypertension, with studies reporting prevalence rates of ~10% in the general hypertensive population and ~20% among patients with resistant hypertension. The cause of primary aldosteronism can be a unilateral aldosterone-producing adenoma (APA) or bilateral idiopathic hyperaldosteronism (IHA) whereby there is diffuse production of ectopic and non-physiologic aldosterone in the adrenal cortex. IHA likely contributes to >70% of all primary aldosteronism. Whereas surgical cure is the preferred therapy for APA, lifelong mineralocorticoid receptor antagonists (MRAs), such as spironolactone or eplerenone, are used to treat IHA. Treatment is important as patients with primary aldosteronism have an elevated risk of adverse cardiovascular and renal outcomes compared to patients with essential hypertension. It was long thought that curative surgery and lifelong medical therapy were equivalent treatment options, but more recent studies suggest that MRAs may not ameliorate the adverse cardiovascular and renovascular effects of primary aldosteronism to the same extent as surgery. For one, MRAs do not lower aldosterone levels, in fact, aldosterone levels are even higher with MRA therapy. Therefore, for IHA patients with primary aldosteronism in whom surgery is not an option, efforts to improve and optimize medical therapy are important.

In recent years, several mutations in cellular membrane ion channels and pumps have been found to cause primary aldosteronism. Nearly all APAs that cause primary aldosteronism harbor an underlying driver mutation in one or more of the following genes: *KCNJ5* (inward-rectifying potassium channel), *ATP1A1* (Na<sup>+</sup>/K<sup>+</sup> ATPase), *ATP2B3* (Ca<sup>2+</sup> ATPase), *CACNA1D* (L-type voltage-dependent Ca<sup>2+</sup> channel), or *CLCN2* (chloride channel). The unifying mechanism of all these gene alterations is that the underlying pathology induces increased calcium ion influx into adrenal zona glomerulosa cells which induces excess aldosterone production.

Moreover, recent evidence in surgically removed adrenal glands from patients with primary aldosteronism and IHA has shown that even though IHA adrenal glands do not harbor adrenal tumors, they do harbor foci of ectopic aldosterone production and these foci are enriched for mutations in *CACNA1D*, thereby suggesting that calcium channel mutations are predominant in the pathogenesis of IHA. This represents an intriguing target for medical therapy as blockade of this channel could lower intracellular calcium and hence decrease aldosterone production. Calcium channel blockade would also represent a more upstream therapy than mineralocorticoid receptor antagonists, which block aldosterone's action at its receptor rather than lower its production.

Calcium channel blockers such as amlodipine are a class of medications that have been used in the treatment of essential hypertension for years and are safe with minimal risks. We hypothesize that amlodipine can lower autonomous aldosterone production in primary aldosteronism patients with IHA, a population that is more likely to harbor a mutation in the L-type voltage-gated calcium channel and a population in whom medical therapy is usually the only treatment option.

# Preliminary Data to Support the Proposed Study

# II. SPECIFIC AIMS

The hypothesis for this **pilot study** is that the calcium-channel blocker amlodipine can specifically decrease aldosterone production in patients with idiopathic bilateral hyperaldosteronism.

- <u>Primary Outcome:</u> Change in 24-hour urinary aldosterone excretion rate and plasma aldosterone in response to maximal amlodipine therapy.
- Secondary Outcomes: Acute change in plasma aldosterone in response to amlodipine therapy.

# III. SUBJECT SELECTION

# Sample Size:

Up to 15 participants with confirmed or presumed IHA will be recruited. Some patients with IHA will have this diagnosis confirmed via adrenal venous sampling. Many patients have not undergone adrenal venous sampling but have a preumptive diagnosis of IHA because they have no adrenal abnormalities on imaging and/or are already being treated with mineralocorticoid receptor antagonists.

Participants will be included if they are aged 18-80 years, have a confirmed diagnosis of primary aldosteronism, a suppressed plasma renin activity (<1.0 ng/mL/h), and confirmed or presumed IHA. Participants taking a calcium-channel blocker will be included if they are willing to undergo a washout protocol (described below). Participants taking mineralocorticoid receptor antagonists will be included if their plasma renin activity is <1.0 ng/mL/h; if it is not, they may still be included if they are able to lower the dose of this medication such that their renin activity falls below 1.0 ng/mL/h.

Participants will be excluded if they have discrete or large bilateral adrenal adenomas on cross-sectional imaging (done as a part of standard clinical care) to avoid including participants who may have APAs, which predominantly have *KCNJ5* mutations rather than *CACNA1D* calcium channel mutations. Participants with anemia, leukopenia, or thrombocytopenia (based on our acceptable ranges) or a blood pressure greater than 180/100 mmHg, will be excluded. Pregnant or breastfeeding women will also be excluded.

# IV. SUBJECT ENROLLMENT

The study will take place at Brigham and Women's Hospital (BWH). Our research team has extensive experience and an established infrastructure for recruiting individuals with IHA. Participants will be recruited from 2 sources.

- Center for Adrenal Disorders at BWH: The PI sees primary aldosteronism patients in the clinic. In addition, participants undergoing adrenal venous sampling for primary aldosteronism will be contacted if they have IHA. Patients with IHA will be contacted regarding interest in participation by the PI's research team with a letter.
- 2. Partners Research Patient Data Registry (RPDR): The Brigham & Women's Hospital and Partners affiliates i.e. Massachusetts General Hospital, Faulkner Hospital, Newton Wellesley, etc. have a shared database to identify potentially eligible patients that can be used for clinical research studies. We will search for patients with primary aldosteronism

in the RPDR and with IRB committee approval, conduct targeted chart reviews to assess which patients likely meet inclusion criteria for this study. Once we have identified potentially eligible patients, they will be invited to participate via the Mass General Brigham Patient Gateway secure online portal or we will identify their primary care physician, or endocrinologist, or other internist with close ties to the patient in our system, and request permission to contact their potentially eligible patient with our IRB approved letter (co-signed by the PI and physician) including information regarding the study. The letter is used to ask permission to send their patients a co-signed letter inviting them to learn more about and potentially participate in our study. In the letter, participants will be notified that we will be calling within about 2 weeks after receipt of the letter. Our phone number will be provided so individuals may contact us with questions or to opt out of receiving further information about the study. Interested patients will be invited for a screening visit to formally assess eligibility.

# V. STUDY PROCEDURES

The study will take place in the outpatient clinical research centers of the BWH. There will be one screening visit, and 3 study visits. The duration of the entire study is 2-10 weeks (see protocol schema).



<u>Screening visit (Visit 1):</u> Participants will meet with a study staff member (licensed physician or nurse practitioner or physician assistant) to review the study protocol, risks, and benefits. They will have received the consent form ahead of this visit and it will be reviewed in detail and signed prior to proceeding. The screening visit will entail a brief review of the patient's medical history, a physical examination, blood pressure measurements, an EKG will be performed, and phlebotomy to assess eligibility. Women between the ages of 18-50 will have a pregnancy test that must be negative.

Blood pressure medication washout and optimization period: Many participants may already be treated with a calcium-channel blocker per standard of care. To assess the effect of amlodipine on aldosterone production, these participants will washout their prescribed calcium-channel blocker for 4-8 weeks and will have their blood pressure managed with other anti-hypertensive agents in the interim. After stopping their calcium-channel blocker, participants will be provided with a home blood pressure machine and taught how to measure their blood pressure at home and how to report daily readings to study staff. The target blood pressure for this washout period, and throughout the entire study protocol, will be 120-150/60-90 mmHg. The upper limit of this blood pressure range exceeds the normal range because many patients with primary aldosteronism have chronically elevated and poorly controlled blood pressure; although study staff will make every effort to maintain their blood pressure in a normal range (<130/80 mmHg),

this goal may not be achievable in this short study. If home blood pressure exceeds 130/80 mmHg, participants will be prescribed doxazosin (in 2 mg daily increments up to 8 mg daily) and/or hydralazine (in 25 mg daily increments up to 25 mg three times daily) in efforts to keep blood pressure in the target range. These medications will be used to substitute calcium-channel blockers since they do not interfere with the renin-angiotensin-aldosterone system and are the recommended medications by the international Endocrine Society guidelines.

In addition to blood pressure monitoring during this washout period, serum potassium will be monitored to ensure it remains in a target range of 3.5-4.5 mEq/L. Most patients with primary aldosteronism are hypokalemic and already taking daily potassium supplements. Study staff may increase the dose of potassium supplementation (using potassium chloride in 20 mEq supplements) to keep serum potassium in the target range. Serum potassium will be checked at 2-4 weeks, and if not in range, again at 4-8 weeks.

Participants already taking a mineralocorticoid receptor antagonist (such as spironolactone or eplerenone) will be included and studied as long as their renin activity remains suppressed (<1.0 ng/mL/h). Participants who have a renin activity greater than or equal to 1.0 ng/mL/h while on mineralocorticoid receptor antagonists may still participate if their dose can be safely decreased such that renin activity decreases to <1.0 ng/mL/h. If needed, renin will be measured at 2-4 weeks, and if not in range, again at 4-8 weeks.

This washout and optimization period will range from 4-8 weeks to provide sufficient time for optimization of washout, blood pressure, potassium, and renin levels. Participants who are unable to tolerate a washout or maintain blood pressure or potassium in the target range, will be withdrawn from the study.

<u>Study Visit 2-Dexamethasone Suppression Test/Cosyntropin stimulation test:</u> After completing the washout period, participants will be scheduled to undergo a dexamethasone suppression test and cosyntropin stimulation test. This will be conducted prior to the high sodium diet given before visit 3.

The dexamethasone suppression test is often used in the clinical setting to measure whether there is excess cortisol secretion. Dexamethasone (1mg) is a synthetic adrenal steroid and is taken the night before the cosyntropin stimulation test between 11pm and 12am. When the participant arrives to the CCI the following morning between 8-9am, initial biochemical testing will include ACTH and cortisol levels. These hormone values will demonstrate how well cortisol can be suppressed.

The cosyntropin stimulation test will measure how well cortisol can be stimulated. A cosyntropin stimulation test is a common procedure that is performed routinely in the ambulatory setting at BWH in the primary care, endocrine, and oncology clinics. It involves the measurement of adrenal hormones before, and one hour after, the administration of cosyntropin (an analogue of the peptide ACTH: "ACTH 1-24"). Participants will arrive to the CCI at 8-9am in the morning and will have an IV placed in the arm. A baseline blood measurement will be analyzed for cortisol, aldosterone, plasma renin activity, direct renin concentration, ACTH, and basic metabolic chemistries. The standard dose of cosyntropin (250 mcg) will then be administered by IV bolus and blood work for cortisol and aldosterone measured again 60mins later. This will conclude the visit which is expected to last ~2hours.

**Study Visits 3 and 4:** Following screening and washout/optimization, there will be two study visits separated by 2 weeks (see Schema Figure). Critical determinants of aldosterone production

include body posture, dietary sodium intake, serum potassium, and blood pressure. Thus, this protocol ensures that all 4 of these confounders are controlled to ensure that outcome measures are reliable and reproducible.

<u>Study Visit 3:</u> The objective for study visit 3 is to establish the magnitude of autonomous aldosterone production at baseline and evaluate the *acute* impact of amlodipine on aldosterone production.

To ensure rigor and reproducibility, all aldosterone (and other measurements) will be conducted under conditions where diet and posture are controlled. Five days before study visit 3, participants will be provided with sodium supplements (in the form of 3 broth packets approximating 3,000 mg of sodium daily) to consume daily. The average daily sodium consumption in the United States is 3.8-4.5 grams daily, and thus this sodium intake will ensure that all participants are consuming a typical U.S. sodium diet and for research purposes, ensure that the 24 hour urinary sodium excretion at study visit 3 is >200 mmol Na<sup>+</sup>/24h. This sodium loading is a standard of care clinical practice referred to as an "oral sodium suppression test" and the internationally recommended test to diagnose primary aldosteronism by the Endocrine Society.

After consuming this sodium diet, participants will arrive at the BWH Clinical Research Center at 8AM, after having collected their urine for 24 hours. An EKG will be performed if the participant had a remote screening visit. Participants will remain in an upright seated position for a total of seven hours. After one hour of seated rest, baseline blood measures will be obtained, and a single dose of amlodipine 10 mg will be administered. In order to reflect amlodipine pharmacodynamics, blood measurements will be repeated every 2 hours to assess the serial change in outcome measures (t=2,4,and 6 hours after the amlodipine dose). This serial blood testing may be performed via repeated venipuncture, or by placing an intravenous line to draw, whichever is preferable to the participant. Blood tests will include serum aldosterone, plasma renin activity, basic metabolic panel, adrenocorticotropic hormone, cortisol, and other hybrid adrenal steroids. Extra plasma and serum will be saved for future use and DNA will be extracted from peripheral leukocytes for genetic analyses of aldosterone-related genes. The 24h urine will be analyzed for aldosterone excretion rate, cortisol, sodium, potassium, and creatinine.

During the study visit, participants will be able to drink water and after a 4-hour period be able to eat a light snack. After the study is completed, participants will be able to eat and encouraged to bring food with them for this.

<u>Treatment phase:</u> Following completion of Visit 3, participants will be prescribed amlodipine 10mg daily for 2 weeks. Home blood pressure monitoring will continue to ensure blood pressure remains in the target range of 120-150/80-90 mmHg. If blood pressure falls below this range with amlodipine, doxazosin and/or hydralazine doses may be reduced or stopped. If blood pressure remains low even after stopping doxazosin and hydralazine, the dose of amlodipine may be lowered to 5mg daily. Potassium chloride supplements may be titrated based on the values obtained at Study visit 3.

<u>Study Visit 4:</u> The objective for study visit 4 is to establish the magnitude of autonomous aldosterone production after 2 weeks of amlodipine treatment.

Participants will again complete 5 days of sodium supplements and arrive to the BWH Clinical Research Center at 8AM, bringing with them a 24-hour urine collection. Participants will be instructed to not take their daily amlodipine dose prior to arriving, they will take it as a part of the study visit. They will repeat the exact same study protocol completed at Visit 3. Participants will

remain in an upright seated position for a total of seven hours. After the first hour of seated rest, baseline blood measures will be obtained and a single dose of amlodipine (the dose will be the same dose they took for the preceding 2 weeks) will be administered. Blood and urinary measurements will again be performed exactly as they were at visit 3.

# VI. BIOSTATISTICAL ANALYSIS

The analytic plan for this pilot study is to compare the change in plasma aldosterone (Aldo) and the change in 24h urinary aldosterone excretion rate (AER). The primary analytic plan will be to evaluate  $\Delta$ Aldo and  $\Delta$ AER between visit 2 and 3. Wilcoxon signed rank, or paired T-test statistics, will be used for univariate statistical analyses to assess significant differences between the paired measurements of  $\Delta$ Aldo and  $\Delta$ AER. Adjustment for potential confounders (age, sex, race/ethnicity, BMI, BP) will be considered using generalized linear mixed random effects models (SAS 9.4). Secondary analyses to assess the acute change in plasma aldosterone after a single dose of amlodipine will be conducted using the same methodological approach.

Sample size calculations are based on an expected  $\triangle Aldo$  of 5 ng/dL, with up to a  $\triangle S.D.$  of 4-5 ng/dL. It is thus estimated that 7-10 participants are needed in this paired design to reject the null hypothesis that  $\triangle Aldo$  does not significantly change with amlodipine therapy with 80% power. Similarly, for an expected  $\triangle AER$  of 7 mcg/24h, with a  $\triangle S.D.$  of 5-6 mcg/24h, it is estimated that 6-8 participants are needed in this paired design to reject the null hypothesis that  $\triangle AER$  does not significantly change with amlodipine therapy with 80% power.

We aim to enroll 15 participants to provide sufficient sample size and power to detect differences even if 2-5 participants (up to 33%) are non-responders to amlodipine. As this is a pilot study, any information regarding the influence of amlodipine on aldosterone production may be useful in designing future studies.

# VII. RISKS AND DISCOMFORTS

### **Sodium supplementation**

The sodium intake is not intrinsically harmful, and in fact contains a similar amount of sodium to the diet consumed by the average American. This sodium intake is also the standard of care, and international guideline recommended approach, to assess aldosterone production in patients with primary aldosteronism. Possible side effects include a rise in blood pressure or drop in serum potassium which study staff will be monitoring closely and will be able to titrate medications to prevent or treat.

### Risk of Washout Period/Risk of Stopping Regular Blood Pressure Medications

During the washout/optimization period, there is a risk that the participants' blood pressure may rise despite initiation of an alternative antihypertensive agent. Risks of high blood pressure include headache and in rare and extreme circumstances stroke, heart attack, and death. Home blood pressure will be closely monitored, and study staff will actively titrate alternative antihypertensive agent(s) to ensure blood pressure remains well-controlled. This is a commonly performed procedure in clinical practice and routine.

### Calcium channel blocker treatment (amlodipine)

Amlodipine is a commonly prescribed medication that has been used to treat essential hypertension for years. The most common side effect is swelling in the legs and ankles (which usually takes 1-2 weeks or longer to manifest). It can also cause low blood pressure particularly at a high dose, but this is unlikely in the current study. Other rare side effects include fluid in the lungs in heart failure patients, palpitations, fatigue, skin rash, and stomach upset.

# Hydralazine

Hydralazine has been used for many years in the treatment of essential hypertension. It is an international guideline recommended medication for treatment in primary aldosteronism when diagnostic testing is conducted. Side effects include low blood pressure, fast heart rate, stomach upset, and headache. Rare side effects include an autoimmune lupus-like syndrome, liver damage, and decreased white blood cell count. It should not be used in patients with coronary artery disease.

### Doxazosin

Doxazosin has been approved for the treatment of essential hypertension for many years. It is an international guideline recommended medication for treatment in primary aldosteronism when diagnostic testing is conducted. Side effects include low blood pressure, leg swelling, nausea, dizziness, and headache. Rare side effects include liver inflammation and angioedema (swelling of the lips and tongue).

### **ACTH infusion**

Cosyntropin is a synthetic derivative of naturally occurring adrenocorticotrophic hormone (ACTH), specifically the first 24 of the 39 amino acids of the hormone. Very rarely, patients with a history of asthma or other forms of allergy may be predisposed to hypersensitivity reaction or anaphylaxis during Cosyntropin administration; bradycardia, tachycardia, hypertension, peripheral edema, and rash have also been reported with cosyntropin. A physician or nurse will be present for the test. This cosyntropin stimulation test is a common ambulatory test that is performed in the clinical setting.

### **Dexamethasone**

Dexamethasone is a synthetic glucocorticoid. Very rarely dexamethasone may cause anaphylactic reactions in those with hypersensitivity to dexamethasone; infection; slow wound healing; diaphoresis; nausea; headache; and mood changes. Most of these reactions are cause from chronic use, not the one-time administration as in our study.

### **Blood Draws/Phlebotomy**

Some may experience a mild sting or painful feeling at the site of needle or intravenous catheter insertion. Although uncommon, it can also lead to a blood clot or infection. Standard sterile precautions will be taken to minimize these risks.

### Pregnancy/Fetus

Women cannot take part in this study if they are pregnant or breastfeeding. Women between the age of 18-50 years will be required to have a negative pregnancy test prior to taking part in the study. Women who are postmenopausal and amenorrheic for one year or who have had a surgical sterilization procedure are exempt from submitting to a pregnancy test. Women will be counseled about using abstinence or contraception during participation in this study to avoid exposure to potentially teratogenic medications.

### **Genetic Information**

Genetic information about this study does not have medical or treatment implications at this time. However, information about participation in a genetic study may influence insurance and/or employers. These risks are minimized by not sharing information about participation and by using de-identified study codes. We will not place genetic information in the medical record. All results and samples will be coded and the key to the code kept in a separate locked file.

In order to allow researchers to share test results, the National Institutes of Health (NIH) and other central repositories have developed special data (information) banks that analyze data and collect the results of whole genome studies. These banks may also analyze and store DNA samples, as well. These central banks will store genetic information and samples and give them to other researchers to do more studies. Although it is impossible to predict how genetic information will be used in the future, there are many safeguards in place to ensure that all genetic information is protected and de-identified.

### **Unknown Risks**

There may be other risks or side effects that are not known at this time.

# VIII. POTENTIAL BENEFITS

Although patients are not expected to directly benefit from the trial, their participation will contribute to medical research. Because of the close monitoring, supervision, and pro-active blood pressure and potassium therapies, participants will likely see an improvement in their primary aldosteronism therapy goals, even though this is not the primary objective of the study.

### IX. REMUNERATION

Patients will receive monetary compensation for participating in the study and parking and/or transportation costs will also be covered. Participants will receive \$100 for completing study visit 3 and \$100 for completing study visit 4. Parking at BWH lots will be covered. For participants who need transportation, reimbursement for public transportation and/or livery services (i.e. Uber, Lyft, taxi, etc) will be strongly considered on a case-by-case basis based on feasibility and location.

# X. MONITORING AND QUALITY ASSURANCE

The Principal Investigator will be responsible for reviewing the safety and/or efficacy data and determining whether the research should be altered or stopped.

Safety data will be reviewed on every case studied in the PI's monthly research group meeting. The PI's research group, the Cardiovascular Endocrinology Research Group (CERG), meets once a month on a Tuesday. The CERG includes more than 5 patient-oriented clinical investigators who are all endocrinologists with detailed knowledge of human research protocols, safety monitoring, and managing hypertension. At each CERG meeting, each PI presents recruitment status, adverse events/safety issues, minor deviations, and other pertinent study-related issues to the group of PI's. Research coordinators also attend this meeting. Discussion of issues and a plan are formulated for each adverse event. The PI will be responsible for executing any plans agreed upon during these meetings.

### REFERENCES

- 1. Rossi GP, Barisa M, Belfiore A, et al. The aldosterone-renin ratio based on the plasma renin activity and the direct renin assay for diagnosing aldosterone-producing adenoma. Journal of hypertension 2010;28:1892-9.
- 2. Mulatero P, Stowasser M, Loh KC, et al. Increased diagnosis of primary aldosteronism, including surgically correctable forms, in centers from five continents. The Journal of clinical endocrinology and metabolism 2004;89:1045-50.
- 3. Funder JW, Carey RM, Fardella C, et al. Case detection, diagnosis, and treatment of patients with primary aldosteronism: an endocrine society clinical practice guideline. The Journal of clinical endocrinology and metabolism 2008;93:3266-81.
- 4. Abdelhamid S, Muller-Lobeck H, Pahl S, et al. Prevalence of adrenal and extra-adrenal Conn syndrome in hypertensive patients. Arch Intern Med 1996;156:1190-5.
- 5. Rossi E, Regolisti G, Negro A, Sani C, Davoli S, Perazzoli F. High prevalence of primary aldosteronism using postcaptopril plasma aldosterone to renin ratio as a screening test among Italian hypertensives. Am J Hypertens 2002;15:896-902.
- 6. Omura M, Saito J, Yamaguchi K, Kakuta Y, Nishikawa T. Prospective study on the prevalence of secondary hypertension among hypertensive patients visiting a general outpatient clinic in Japan. Hypertension research: official journal of the Japanese Society of Hypertension 2004;27:193-202.
- 7. Rossi GP, Bernini G, Caliumi C, et al. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. Journal of the American College of Cardiology 2006;48:2293-300.
- 8. Fogari R, Preti P, Zoppi A, Rinaldi A, Fogari E, Mugellini A. Prevalence of primary aldosteronism among unselected hypertensive patients: a prospective study based on the use of an aldosterone/renin ratio above 25 as a screening test. Hypertens Res 2007;30:111-7.
- 9. Hannemann A, Bidlingmaier M, Friedrich N, et al. Screening for primary aldosteronism in hypertensive subjects: results from two German epidemiological studies. European journal of endocrinology / European Federation of Endocrine Societies 2012;167:7-15.
- 10. Sang X, Jiang Y, Wang W, et al. Prevalence of and risk factors for primary aldosteronism among patients with resistant hypertension in China. Journal of hypertension 2013;31:1465-71; discussion 71-2.
- 11. Monticone S, Burrello J, Tizzani D, et al. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. Journal of the American College of Cardiology 2017;69:1811-20.
- 12. Lim PO, Dow E, Brennan G, Jung RT, MacDonald TM. High prevalence of primary aldosteronism in the Tayside hypertension clinic population. Journal of human hypertension 2000;14:311-5.
- 13. Gordon RD, Stowasser M, Tunny TJ, Klemm SA, Rutherford JC. High incidence of primary aldosteronism in 199 patients referred with hypertension. Clinical and experimental pharmacology & physiology 1994;21:315-8.
- 14. Gallay BJ, Ahmad S, Xu L, Toivola B, Davidson RC. Screening for primary aldosteronism without discontinuing hypertensive medications: plasma aldosterone-renin ratio. American journal of kidney diseases: the official journal of the National Kidney Foundation 2001;37:699-705.
- 15. Williams D, Croal B, Furnace J, et al. The prevalence of a raised aldosterone-renin ratio (ARR) among new referrals to a hypertension clinic. Blood Press 2006;15:164-8.
- 16. Williams JS, Williams GH, Raji A, et al. Prevalence of primary hyperaldosteronism in mild to moderate hypertension without hypokalaemia. J Hum Hypertens 2006;20:129-36.
- 17. Westerdahl C, Bergenfelz A, Isaksson A, Wihl A, Nerbrand C, Valdemarsson S. High frequency of primary hyperaldosteronism among hypertensive patients from a primary care area in Sweden. Scand J Prim Health Care 2006;24:154-9.

- 18. Calhoun DA, Nishizaka MK, Zaman MA, Thakkar RB, Weissmann P. Hyperaldosteronism among black and white subjects with resistant hypertension. Hypertension 2002;40:892-6.
- 19. Benchetrit S, Bernheim J, Podjarny E. Normokalemic hyperaldosteronism in patients with resistant hypertension. Isr Med Assoc J 2002;4:17-20.
- 20. Douma S, Petidis K, Doumas M, et al. Prevalence of primary hyperaldosteronism in resistant hypertension: a retrospective observational study. Lancet 2008;371:1921-6.
- 21. Nogueira AR, Bloch KV. Screening for primary aldosteronism in a cohort of Brazilian patients with resistant hypertension. J Clin Hypertens (Greenwich) 2008;10:619-23.
- 22. Ribeiro MJ, Figueiredo Neto JA, Memoria EV, et al. Prevalence of primary hyperaldosteronism in a systemic arterial hypertension league. Arq Bras Cardiol 2009;92:39-45.
- 23. Monticone S, D'Ascenzo F, Moretti C, et al. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. The lancet Diabetes & endocrinology 2018;6:41-50.
- 24. Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Cardiometabolic outcomes and mortality in medically treated primary aldosteronism: a retrospective cohort study. The lancet Diabetes & endocrinology 2018;6:51-9.
- 25. Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Incidence of Atrial Fibrillation and Mineralocorticoid Receptor Activity in Patients With Medically and Surgically Treated Primary Aldosteronism. JAMA cardiology 2018;3:768-74.
- 26. Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Renal Outcomes in Medically and Surgically Treated Primary Aldosteronism. Hypertension 2018;72:658-66.
- 27. Rossi GP, Bernini G, Desideri G, et al. Renal damage in primary aldosteronism: results of the primary aldosteronismPY Study. Hypertension 2006;48:232-8.
- 28. Reincke M, Rump LC, Quinkler M, et al. Risk factors associated with a low glomerular filtration rate in primary aldosteronism. The Journal of clinical endocrinology and metabolism 2009:94:869-75.
- 29. Hundemer GL, Baudrand R, Brown JM, Curhan G, Williams GH, Vaidya A. Renin Phenotypes Characterize Vascular Disease, Autonomous Aldosteronism, and Mineralocorticoid Receptor Activity. The Journal of clinical endocrinology and metabolism 2017;102:1835-43.
- 30. Sechi LA, Novello M, Lapenna R, et al. Long-term renal outcomes in patients with primary aldosteronism. Jama 2006;295:2638-45.
- 31. Funder JW. Primary aldosteronism: clinical lateralization and costs. The Journal of clinical endocrinology and metabolism 2012;97:3450-2.
- 32. Kupers EM, Amar L, Raynaud A, Plouin PF, Steichen O. A clinical prediction score to diagnose unilateral primary aldosteronism. The Journal of clinical endocrinology and metabolism 2012;97:3530-7.
- 33. Calhoun DA. Is there an unrecognized epidemic of primary aldosteronism? Pro. Hypertension 2007;50:447-53; discussion -53.
- 34. Young MJ. Targeting the mineralocorticoid receptor in cardiovascular disease. Expert Opin Ther Targets 2013;17:321-31.
- 35. Funder JW. Mineralocorticoid receptor antagonists: emerging roles in cardiovascular medicine. Integrated blood pressure control 2013;6:129-38.
- 36. Ma TK, Szeto CC. Mineralocorticoid receptor antagonist for renal protection. Renal failure 2012;34:810-7.
- 37. Brown NJ. Contribution of aldosterone to cardiovascular and renal inflammation and fibrosis. Nat Rev Nephrol 2013;9:459-69.
- 38. Gilbert KC, Brown NJ. Aldosterone and inflammation. Current opinion in endocrinology, diabetes, and obesity 2010;17:199-204.

- 39. Carey RM. Aldosterone and cardiovascular disease. Current opinion in endocrinology, diabetes, and obesity 2010;17:194-8.
- 40. Freel EM, Mark PB, Weir RA, et al. Demonstration of blood pressure-independent noninfarct myocardial fibrosis in primary aldosteronism: a cardiac magnetic resonance imaging study. Circ Cardiovasc Imaging 2012;5:740-7.
- 41. Stehr CB, Mellado R, Ocaranza MP, et al. Increased levels of oxidative stress, subclinical inflammation, and myocardial fibrosis markers in primary aldosteronism patients. Journal of hypertension 2010;28:2120-6.
- 42. Zhou X, Ono H, Ono Y, Frohlich ED. Aldosterone antagonism ameliorates proteinuria and nephrosclerosis independent of glomerular dynamics in L-NAME/SHR model. American journal of nephrology 2004;24:242-9.
- 43. Savard S, Amar L, Plouin PF, Steichen O. Cardiovascular complications associated with primary aldosteronism: a controlled cross-sectional study. Hypertension 2013;62:331-6.
- 44. Milan A, Magnino C, Fabbri A, et al. Left heart morphology and function in primary aldosteronism. High blood pressure & cardiovascular prevention: the official journal of the Italian Society of Hypertension 2012;19:11-7.
- 45. Mulatero P, Monticone S, Bertello C, et al. Long-term cardio- and cerebrovascular events in patients with primary aldosteronism. The Journal of clinical endocrinology and metabolism 2013;98:4826-33.
- 46. Young WF, Jr. Minireview: primary aldosteronism--changing concepts in diagnosis and treatment. Endocrinology 2003;144:2208-13.
- 47. Choi M, Scholl UI, Yue P, et al. K+ channel mutations in adrenal aldosterone-producing adenomas and hereditary hypertension. Science 2011;331:768-72.
- 48. Beuschlein F, Boulkroun S, Osswald A, et al. Somatic mutations in ATP1A1 and ATP2B3 lead to aldosterone-producing adenomas and secondary hypertension. Nature genetics 2013;45:440-4, 4e1-2.
- 49. Azizan EAB, Poulsen H, Tuluc P, et al. Somatic mutations in ATP1A1 and CACNA1D underlie a common subtype of adrenal hypertension. Nature genetics 2013;45:1055-60. 50. Scholl UI, Goh G, Stolting G, et al. Somatic and germline CACNA1D calcium channel mutations in aldosterone-producing adenomas and primary aldosteronism. Nature genetics
- 2013;45:1050-4. 51. Scholl UI, Stolting G, Nelson-Williams C, et al. Recurrent gain of function mutation in calcium channel CACNA1H causes early-onset hypertension with primary aldosteronism.
- 52. Scholl UI, Stolting G, Schewe J, et al. CLCN2 chloride channel mutations in familial hyperaldosteronism type II. Nature genetics 2018.

eLife 2015;4:e06315.

- 53. Fernandes-Rosa FL, Daniil G, Orozco IJ, et al. A gain-of-function mutation in the CLCN2 chloride channel gene causes primary aldosteronism. Nature genetics 2018.
- 54. Monticone S, Hattangady NG, Nishimoto K, et al. Effect of KCNJ5 mutations on gene expression in aldosterone-producing adenomas and adrenocortical cells. The Journal of clinical endocrinology and metabolism 2012;97:E1567-72.
- 55. Monticone S, Hattangady NG, Penton D, et al. a Novel Y152C KCNJ5 mutation responsible for familial hyperaldosteronism type III. The Journal of clinical endocrinology and metabolism 2013;98:E1861-5.
- 56. Oki K, Plonczynski MW, Luis Lam M, Gomez-Sanchez EP, Gomez-Sanchez CE. Potassium channel mutant KCNJ5 T158A expression in HAC-15 cells increases aldosterone synthesis. Endocrinology 2012;153:1774-82.
- 57. Williams TA, Monticone S, Schack VR, et al. Somatic ATP1A1, ATP2B3, and KCNJ5 Mutations in Aldosterone-Producing Adenomas. Hypertension 2014;63:188-95.

- 58. Tauber P, Aichinger B, Christ C, et al. Cellular Pathophysiology of an Adrenal Adenoma-Associated Mutant of the Plasma Membrane Ca(2+)-ATPase ATP2B3. Endocrinology 2016;157:2489-99.
- 59. Fernandes-Rosa FL, Williams TA, Riester A, et al. Genetic spectrum and clinical correlates of somatic mutations in aldosterone-producing adenoma. Hypertension 2014;64:354-61.
- 60. Sasano H. Localization of steroidogenic enzymes in adrenal cortex and its disorders. Endocrine journal 1994;41:471-82.
- 61. Omata K, Satoh F, Morimoto R, et al. Cellular and Genetic Causes of Idiopathic Hyperaldosteronism. Hypertension 2018;72:874-80.
- 62. Nanba K, Chen AX, Omata K, et al. Molecular Heterogeneity in Aldosterone-Producing Adenomas. The Journal of clinical endocrinology and metabolism 2016;101:999-1007.
- 63. Hattangady NG, Karashima S, Yuan L, et al. Mutated KCNJ5 activates the acute and chronic regulatory steps in aldosterone production. Journal of molecular endocrinology 2016:57:1-11.
- 64. Nanba K, Omata K, Tomlins SA, et al. Double adrenocortical adenomas harboring independent KCNJ5 and PRKACA somatic mutations. Eur J Endocrinol 2016;175:K1-6.
- 65. Omata K, Yamazaki Y, Nakamura Y, et al. Genetic and Histopathologic Intertumor Heterogeneity in Primary Aldosteronism. J Clin Endocrinol Metab 2017;102:1792-6.
- 66. Yamazaki Y, Nakamura Y, Omata K, et al. Histopathological Classification of Cross-Sectional Image-Negative Hyperaldosteronism. The Journal of clinical endocrinology and metabolism 2017;102:1182-92.
- 67. Nanba AT, Nanba K, Byrd JB, et al. Discordance between imaging and immunohistochemistry in unilateral primary aldosteronism. Clinical endocrinology 2017;87:665-72.
- 68. Nanba K, Omata K, Else T, et al. Targeted Molecular Characterization of Aldosterone-Producing Adenomas in White Americans. J Clin Endocrinol Metab 2018;103:3869-76.
- 69. Nanba K, Omata K, Gomez-Sanchez CE, et al. Genetic Characteristics of Aldosterone-Producing Adenomas in Blacks. Hypertension 2019:HYPERTENSIONAHA11812070.
- 70. Lerario AM, Nanba K, Blinder AR, et al. Genetics of aldosterone-producing adenomas with pathogenic KCNJ5 variants. Endocrine-related cancer 2019.
- 71. Nanba K, Vaidya A, Williams GH, Zheng I, Else T, Rainey WE. Age-Related Autonomous Aldosteronism. Circulation 2017;136:347-55.
- 72. Omata K, Anand SK, Hovelson DH, et al. Aldosterone-Producing Cell Clusters Frequently Harbor Somatic Mutations and Accumulate With Age in Normal Adrenals. J Endocr Soc 2017;1:787-99.
- 73. Sun N, Wu Y, Nanba K, et al. High-Resolution Tissue Mass Spectrometry Imaging Reveals a Refined Functional Anatomy of the Human Adult Adrenal Gland. Endocrinology 2018;159:1511-24.
- 74. Omata K, Tomlins SA, Rainey WE. Aldosterone-Producing Cell Clusters in Normal and Pathological States. Horm Metab Res 2017;49:951-6.
- 75. Nanba K, Vaidya A, Rainey WE. Aging and Adrenal Aldosterone Production. Hypertension 2018;71:218-23.
- 76. Mulatero P, Tauber P, Zennaro MC, et al. KCNJ5 mutations in European families with nonglucocorticoid remediable familial hyperaldosteronism. Hypertension 2012;59:235-40.
- 77. Meyer LS, Wang X, Susnik E, et al. Immunohistopathology and Steroid Profiles Associated With Biochemical Outcomes After Adrenalectomy for Unilateral Primary Aldosteronism. Hypertension 2018;72:650-7.
- 78. Stindl J, Tauber P, Sterner C, Tegtmeier I, Warth R, Bandulik S. Pathogenesis of Adrenal Aldosterone-Producing Adenomas Carrying Mutations of the Na(+)/K(+)-ATPase. Endocrinology 2015;156:4582-91.

- 79. Xie CB, Shaikh LH, Garg S, et al. Regulation of aldosterone secretion by Cav1.3. Scientific reports 2016;6:24697.
- 80. Wang T, Satoh F, Morimoto R, et al. Gene expression profiles in aldosterone-producing adenomas and adjacent adrenal glands. European journal of endocrinology / European Federation of Endocrine Societies 2011;164:613-9.
- 81. Nogueira EF, Gerry D, Mantero F, Mariniello B, Rainey WE. The role of TASK1 in aldosterone production and its expression in normal adrenal and aldosterone-producing adenomas. Clinical endocrinology 2010;73:22-9.
- 82. Bassett MH, Mayhew B, Rehman K, et al. Expression profiles for steroidogenic enzymes in adrenocortical disease. The Journal of clinical endocrinology and metabolism 2005;90:5446-55.
- 83. Felizola SJ, Nakamura Y, Ono Y, et al. PCP4: a regulator of aldosterone synthesis in human adrenocortical tissues. Journal of molecular endocrinology 2014.
- 84. Bird IM, Hanley NA, Word RA, et al. Human NCI-H295 adrenocortical carcinoma cells: a model for angiotensin-II-responsive aldosterone secretion. Endocrinology 1993;133:1555-61.
- 85. Rainey WE, Bird IM, Mason JI. The NCI-H295 cell line: a pluripotent model for human adrenocortical studies. Molecular and cellular endocrinology 1994;100:45-50.
- 86. Wang T, Rowland JG, Parmar J, Nesterova M, Seki T, Rainey WE. Comparison of aldosterone production among human adrenocortical cell lines. Hormone and metabolic research = Hormon- und Stoffwechselforschung = Hormones et metabolisme 2012;44:245-50.
- 87. Xing Y, Parker CR, Edwards M, Rainey WE. ACTH is a potent regulator of gene expression in human adrenal cells. Journal of molecular endocrinology 2010;45:59-68.
- 88. Xing Y, Edwards MA, Ahlem C, et al. The effects of ACTH on steroid metabolomic profiles in human adrenal cells. The Journal of endocrinology 2011;209:327-35.
- 89. Xing Y, Rainey WE, Apolzan JW, Francone OL, Harris RB, Bollag WB. Adrenal cell aldosterone production is stimulated by very-low-density lipoprotein (VLDL). Endocrinology 2012;153:721-31.
- 90. Bassett MH, Suzuki T, Sasano H, White PC, Rainey WE. The orphan nuclear receptors NURR1 and NGFIB regulate adrenal aldosterone production. Molecular endocrinology 2004;18:279-90.
- 91. Bassett MH, White PC, Rainey WE. A role for the NGFI-B family in adrenal zonation and adrenocortical disease. Endocrine research 2004;30:567-74.
- 92. Bassett MH, White PC, Rainey WE. The regulation of aldosterone synthase expression. Molecular and cellular endocrinology 2004;217:67-74.
- 93. Clyne CD, Nguyen A, Rainey WE. The effects of KN62, a Ca2+/calmodulin-dependent protein kinase II inhibitor, on adrenocortical cell aldosterone production. Endocrine research 1995;21:259-65.
- 94. Clyne CD, White PC, Rainey WE. Calcium regulates human CYP11B2 transcription. Endocrine research 1996;22:485-92.
- 95. Clyne CD, Zhang Y, Slutsker L, Mathis JM, White PC, Rainey WE. Angiotensin II and potassium regulate human CYP11B2 transcription through common cis-elements. Molecular endocrinology 1997;11:638-49.
- 96. Condon JC, Pezzi V, Drummond BM, Yin S, Rainey WE. Calmodulin-dependent kinase I regulates adrenal cell expression of aldosterone synthase. Endocrinology 2002;143:3651-7. 97. Hattangady NG, Olala LO, Bollag WB, Rainey WE. Acute and chronic regulation of aldosterone production. Molecular and cellular endocrinology 2012;350:151-62.
- 98. Nogueira EF, Rainey WE. Regulation of aldosterone synthase by activator transcription factor/cAMP response element-binding protein family members. Endocrinology 2010;151:1060-70.

- 99. Nogueira EF, Vargas CA, Otis M, Gallo-Payet N, Bollag WB, Rainey WE. Angiotensin-II acute regulation of rapid response genes in human, bovine, and rat adrenocortical cells. J Mol Endocrinol 2007;39:365-74.
- 100. Nogueira EF, Xing Y, Morris CA, Rainey WE. Role of angiotensin II-induced rapid response genes in the regulation of enzymes needed for aldosterone synthesis. Journal of molecular endocrinology 2009;42:319-30.
- 101. Pezzi V, Clark BJ, Ando S, Stocco DM, Rainey WE. Role of calmodulin-dependent protein kinase II in the acute stimulation of aldosterone production. The Journal of steroid biochemistry and molecular biology 1996;58:417-24.
- 102. Pezzi V, Clyne CD, Ando S, Mathis JM, Rainey WE. Ca(2+)-regulated expression of aldosterone synthase is mediated by calmodulin and calmodulin-dependent protein kinases. Endocrinology 1997;138:835-8.
- 103. Kumar-Sinha C, Chinnaiyan AM. Precision oncology in the age of integrative genomics. Nature biotechnology 2018;36:46-60.
- 104. Zheng S, Cherniack AD, Dewal N, et al. Comprehensive Pan-Genomic Characterization of Adrenocortical Carcinoma. Cancer cell 2016;29:723-36.
- 105. Rege J, Nishimoto HK, Nishimoto K, Rodgers RJ, Auchus RJ, Rainey WE. Bone Morphogenetic Protein-4 (BMP4): A Paracrine Regulator of Human Adrenal C19 Steroid Synthesis. Endocrinology 2015;156:2530-40.
- 106. Rege J, Karashima S, Lerario AM, et al. Age-dependent Increases in Adrenal Cytochrome b5 and Serum 5-Androstenediol-3-sulfate. The Journal of clinical endocrinology and metabolism 2016;101:4585-93.
- 107. Nakamura Y, Rege J, Satoh F, et al. Liquid chromatography-tandem mass spectrometry analysis of human adrenal vein corticosteroids before and after adrenocorticotropic hormone stimulation. Clinical endocrinology 2012;76:778-84.
- 108. Tauber P, Penton D, Stindl J, et al. Pharmacology and pathophysiology of mutated KCNJ5 found in adrenal aldosterone-producing adenomas. Endocrinology 2014;155:1353-62.
- 109. Funder JW, Carey RM, Mantero F, et al. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. The Journal of clinical endocrinology and metabolism 2016;101:jc20154061.
- 110. Vaidya A, Malchoff CD, Auchus RJ, Committee AAS. An Individualized Approach to the Evaluation and Management of Primary Aldosteronism. Endocr Pract 2017;23:680-9.
- 111. Hundemer G, Curhan G, Yozamp N, Wang M, Vaidya A. Incidence of Atrial Fibrillation and Mineralocorticoid Receptor Activity in Patients with Medically and Surgically Treated Primary Aldosteronism. JAMA Cardiology 2018;**3**:768-74.
- Hundemer G, Curhan G, Yozamp N, Wang M, Vaidya A. Renal Outcomes in Medically Treated Primary Aldosteronism. Hypertension 2018;**72**:658-66.
- 113. Wu VC, Chueh SJ, Chen L, et al. Risk of new-onset diabetes mellitus in primary aldosteronism: a population study over 5 years. J Hypertens 2017;35:1698-708.
- 114. Wu VC, Wang SM, Chang CH, et al. Long term outcome of Aldosteronism after target treatments. Sci Rep 2016;6:32103.
- 115. Omata K, Satoh F, Morimoto R, et al. Cellular and Genetic Causes of Idiopathic Hyperaldosteronism. Hypertension 2018;in press, epub ahead of print.
- 116. Kline GA, Darras P, Leung AA, So B, Chin A, Holmes DT. Surprisingly low aldosterone levels in peripheral veins following intravenous sedation during adrenal vein sampling: implications for the concept of nonsuppressibility in primary aldosteronism. J Hypertens 2019;37:596-602.

- 117. Kowarski A, de Lacerda L, Migeon CJ. Integrated concentration of plasma aldosterone in normal subjects: correlation with cortisol. J Clin Endocrinol Metab 1975;40:205-10.
- 118. Nadler JL, Hsueh W, Horton R. Therapeutic effect of calcium channel blockade in primary aldosteronism. J Clin Endocrinol Metab 1985;60:896-9.